CLINICAL TRIAL: NCT03873584
Title: Multi-center, Non-interventional, Prospective, Clinical Observational Study to Evaluate the Efficacy of Iron Protein Succinylate in Improving Fatigue Symptoms in Patients With Iron Deficiency Anemia
Brief Title: Improvement of Fatigue Symptoms in the Iron Deficiency Anemia With Iron Succinylate Therapy
Acronym: IFAISTOS
Status: Withdrawn | Type: Observational
Why Stopped: no patients enrolment
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-IRPS-EL-99
Record Dates: First submitted 2019-03-12; First posted 2019-03-13 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Anemia; Iron-deficiency; Iron Deficiency Anemia; Fatigue
MeSH Terms: conditions — Anemia; Anemia, Iron-Deficiency; Fatigue

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Fatigue — Iron deficiency anemia with fatigue symptoms

SUMMARY:
The treatment of anemia depends on its cause. Patients with underlying iron-deficient anemia should be treated or referred to a specialist (eg gynecologist, gastroenterologist) for treatment.deficiency anemia are global health problems and common medical conditions seen in everyday clinical practice.

Iron is vital for biological functions, such as breathing, energy production, DNA synthesis, and cell proliferation.

Iron deficiency refers to the reduction of iron stores and precedes the occurrence of iron deficiency anemia.

Iron deficiency anemia is a more severe condition in which low levels of iron are associated with anemia and the presence of small cellular red blood cells.

DETAILED DESCRIPTION:
The diagnosis of anemia is based on the patient's symptoms and blood tests. Blood tests refer to hemoglobin, hematocrit, and the number of red blood cells (per cubic centimeter or millet of blood). Also, the status of iron stores in the body can be measured by measuring ferritin. With these blood tests it can be determined Per os treatment: The dosage of elemental iron required to treat anemia due to iron deficiency in adults is 120 mg per day for three months. An increase in hemoglobin by 1g / dl after one month of treatment shows an adequate response to treatment and confirms the diagnosis. In adults, treatment should be continued for three months after correction of anemia to allow replenishment of iron stores.

Patient noncompliance may be an obstacle to oral therapy due to the occurrence of gastrointestinal side effects such as epigastric discomfort, nausea, diarrhea and constipation. These effects can be reduced when iron is taken with meals but its absorption can be reduced by 40%.

In addition, taking medications such as proton pump inhibitors and agents that reduce gastric acid hypersecretion (eg chronic atrophic gastritis, recent gastrectomy or abdominal incision) reduce iron absorption.

ELIGIBILITY:
Inclusion Criteria:

* 16-90 yers
* Iron deficiency anemia
* Treatment with iron succinylate
* Fatigue symptoms
* Informed Consent
* Compliance with study procedures

Exclusion Criteria:

* Anemia caused by other parameters (non-iron-deficiency)

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 2400 iron deficient patients with fatigue symptoms who are treated with iron succinylate.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Fatigue Symptoms in Iron Deficiency Anaemia | 3 months
  Fatigue Assessment Scale (FAS) rating

SECONDARY OUTCOMES:
Hemoglobin levels | 3 months
  Evaluation of iron succinylate treatment in improving hematological parameters

IPD SHARING:
Plan to Share IPD: Undecided